CLINICAL TRIAL: NCT00079274
Title: A Randomized Phase III Trial of Oxaliplatin (OXAL) Plus 5-Fluorouracil (5-FU)/Leucovorin (CF) With or Without Cetuximab (C225) After Curative Resection for Patients With Stage III Colon Cancer
Brief Title: Comparison of Combination Chemotherapy Regimens With or Without Cetuximab in Treating Patients Who Have Undergone Surgery For Stage III Colon Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Eastern Cooperative Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00639; N0147; U10CA025224 (NIH); CDR0000355132 (Registry Identifier: PDQ (Physician Data Query)); NCT00170092 (obsolete NCT alias)
Record Dates: First submitted 2004-03-08; First posted 2004-03-10 (Estimated); Results first posted 2015-02-09 (Estimated); Last update posted 2020-05-13 (Actual); Status verified 2020-04

CONDITIONS: Adenocarcinoma of the Colon; Stage III Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Irinotecan; Oxaliplatin; Leucovorin; Fluorouracil; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Arm A (combination chemotherapy) (Experimental): Patients received oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, and fluorouracil IV continuously over 46-48 hours on days 1. Treatment repeated every 14 days for up to 12 courses in the absence of unacceptable toxicity or recurrent disease.
  Interventions: Drug: oxaliplatin; Drug: leucovorin calcium; Drug: fluorouracil
- Arm B (combination chemotherapy) (Experimental): Patients received irinotecan IV over 2 hours on day 1 and leucovorin calcium and fluorouracil as in arm A. Treatment repeated every 14 days for up to 12 courses in the absence of unacceptable toxicity or recurrent disease.
  Interventions: Drug: irinotecan hydrochloride; Drug: leucovorin calcium; Drug: fluorouracil
- Arm C (combination chemotherapy) (Experimental): Patients received the same treatment as in arm A for 6 courses followed by the same treatment as in arm B for 6 courses (total of 12 courses). Treatment continues in the absence of unacceptable toxicity or recurrent disease.
  Interventions: Drug: irinotecan hydrochloride; Drug: oxaliplatin; Drug: leucovorin calcium; Drug: fluorouracil
- Arm D (combination chemotherapy, monoclonal antibody) (Experimental): Patients received cetuximab IV over 1 hour on days 1 and 8 and oxaliplatin, leucovorin calcium, and fluorouracil as in arm A. Treatment repeated every 14 days for up to 12 courses in the absence of unacceptable toxicity or recurrent disease.
  Interventions: Drug: oxaliplatin; Drug: leucovorin calcium; Drug: fluorouracil; Biological: cetuximab
- Arm E (combination chemotherapy, monoclonal antibody) (Experimental): Patients received cetuximab as in arm D and irinotecan, leucovorin calcium, and fluorouracil as in arm B. Treatment repeated every 14 days for up to 12 courses in the absence of unacceptable toxicity or recurrent disease.
  Interventions: Drug: irinotecan hydrochloride; Drug: leucovorin calcium; Drug: fluorouracil; Biological: cetuximab
- Arm F (combination chemotherapy, monoclonal antibody) (Experimental): Patients received cetuximab as in arm D and chemotherapy as in arm C.
  Interventions: Drug: irinotecan hydrochloride; Drug: oxaliplatin; Drug: leucovorin calcium; Drug: fluorouracil; Biological: cetuximab
- Arm G (Locally directed therapy) (Other): Patients determined to have mutated KRAS (or KRAS not evaluable) were assigned to an event monitoring arm in which adjuvant therapy was determined and assigned by the treating oncologist. The determination of the type of therapy, duration of treatment, and dose modification was the responsibility of the treating oncologists.
  Interventions: Drug: Locally Directed Therapy

INTERVENTIONS:
Drug: irinotecan hydrochloride — Given IV
  Other Names: Campto; Camptosar; CPT-11; irinotecan; U-101440E
  Arms: Arm B (combination chemotherapy); Arm C (combination chemotherapy); Arm E (combination chemotherapy, monoclonal antibody); Arm F (combination chemotherapy, monoclonal antibody)
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
  Arms: Arm A (combination chemotherapy); Arm C (combination chemotherapy); Arm D (combination chemotherapy, monoclonal antibody); Arm F (combination chemotherapy, monoclonal antibody)
Drug: leucovorin calcium — Given IV
  Other Names: CF; CFR; LV
  Arms: Arm A (combination chemotherapy); Arm B (combination chemotherapy); Arm C (combination chemotherapy); Arm D (combination chemotherapy, monoclonal antibody); Arm E (combination chemotherapy, monoclonal antibody); Arm F (combination chemotherapy, monoclonal antibody)
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
  Arms: Arm A (combination chemotherapy); Arm B (combination chemotherapy); Arm C (combination chemotherapy); Arm D (combination chemotherapy, monoclonal antibody); Arm E (combination chemotherapy, monoclonal antibody); Arm F (combination chemotherapy, monoclonal antibody)
Biological: cetuximab — Given IV
  Other Names: C225; C225 monoclonal antibody; IMC-C225; MOAB C225; monoclonal antibody C225
  Arms: Arm D (combination chemotherapy, monoclonal antibody); Arm E (combination chemotherapy, monoclonal antibody); Arm F (combination chemotherapy, monoclonal antibody)
Drug: Locally Directed Therapy — Patients determined to have mutated KRAS (or KRAS not evaluable) will be assigned to an event monitoring arm in which adjuvant therapy will be determined and assigned by the treating oncologist. The determination of the type of therapy, duration of treatment, and dose modification will be the responsibility of the treating oncologists.
  Arms: Arm G (Locally directed therapy)

SUMMARY:
This randomized phase III trial was originally designed to compare three different combination chemotherapy regimens to see how well they work. As of September 1, 2004, the study was expanded to a total of 6 arms (the original 3 arms (A, B, C) and 3 additional arms which were the same as the first 3 but with cetuximab) in treating patients who have undergone surgery for stage III colon cancer. Drugs used in chemotherapy, such as irinotecan hydrochloride, fluorouracil, leucovorin calcium, and oxaliplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies such as cetuximab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Combining more than one chemotherapy drug with monoclonal antibody therapy and giving them after surgery may kill any remaining tumor cells. It was not known at the time this study was developed which combination chemotherapy regimen is more effective after surgery in treating colon cancer. This study had several key changes, based on the results of other phase III trials. As of 6/1/2005, patients no longer received irinotecan on this study and treatment arms B, C, E, and F were discontinued. Patients on arms B and C crossed to arm A. Patients on arms E and F crossed to arm D. Patients on arms C and F who had not gotten to irinotecan continued on arms A and D, respectively. As of 8/18/2008, pre-screening for Kirsten rat sarcoma (KRAS) status was added with mutant KRAS (or KRAS not evaluable) patients put on arm G and wild-type KRAS patients randomized between arm A and arm D. Patients on arm G were treated per physician discretion and followed for disease and survival status. KRAS was determined in a central laboratory and was process for all patients on this study. The primary endpoint of this study was modified on 8/18/2008 to focus on patients having wild-type KRAS tumors. All modifications were approved by the Central Institution Review Board, local Institutional Review Boards, NCI, and the NCCTG Data Safety Monitoring Board.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Disease-free Survival (Arms A and D: Wild-type KRAS Patients)

SECONDARY OBJECTIVES:

I. Disease-free Survival (Arms A and D: Mutant KRAS Patients) II. Disease-free Survival III. Overall Survival IV. Toxicity

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to positive lymph node involvement (1-3 vs 4 or more), histology (high [poorly differentiated or undifferentiated] vs low [well to moderately differentiated]), and clinical T stage (T1 or T2 vs T3 vs T4). Patients are randomized to 1 of 6 treatment arms (as of 6/1/2005, patients are randomized to treatment arms I and IV only; arms II, III, V, and VI are closed to accrual). As of 8/18/2008, pre-screening for KRAS status was added with mutant KRAS (or KRAS not evaluable) patients put on arm G and wild-type KRAS patients randomized between arm A and arm D.

ARM A: Patients receive oxaliplatin intravenously (IV) over 2 hours, leucovorin calcium IV over 2 hours, and fluorouracil IV continuously over 46-48 hours on days 1. Treatment repeats every 14 days for up to 12 courses in the absence of unacceptable toxicity or recurrent disease.

ARM B (closed to accrual as of 6/1/2005--currently enrolled patients may cross over to arm I for remainder of therapy): Patients receive irinotecan hydrochloride IV over 2 hours on day 1 and leucovorin calcium and fluorouracil as in arm A. Treatment repeats every 14 days for up to 12 courses in the absence of unacceptable toxicity or recurrent disease.

ARM C (closed to accrual as of 6/1/2005--currently enrolled patients may cross over to arm I for remainder of therapy): Patients receive the same treatment as in arm A for 6 courses followed by the same treatment as in arm B for 6 courses (total of 12 courses). Treatment continues in the absence of unacceptable toxicity or recurrent disease.

ARM D: Patients receive cetuximab* IV over 1 hour on days 1 and 8 and oxaliplatin, leucovorin calcium, and fluorouracil as in arm A. Treatment repeats every 14 days for up to 12 courses in the absence of unacceptable toxicity or recurrent disease.

ARM E (closed to accrual as of 6/1/2005--currently enrolled patients may cross over to arm D for remainder of therapy): Patients receive cetuximab* as in arm D and irinotecan hydrochloride, leucovorin calcium, and fluorouracil as in arm B. Treatment repeats every 14 days for up to 12 courses in the absence of unacceptable toxicity or recurrent disease.

ARM F (closed to accrual as of 6/1/2005--currently enrolled patients may cross over to arm D for remainder of therapy): Patients receive cetuximab* as in arm D and chemotherapy as in arm C.

ARM G (added as of 8/18/2008, mutant KRAS (or KRAS not evaluable) patients): Locally directed therapy.

NOTE: *Cetuximab is administered over 2 hours at a higher dose on day 1 of course 1 only.

Quality of life (QOL) is assessed at baseline, 3 months, and at the end of therapy. As of 8/18/2008, QOL was discontinued.

Patients are followed for a maximum of 8 years from randomization.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the colon

  * Stage III disease
  * No resected stage IV disease
* No rectal cancer

  * Gross inferior (caudad) margin of the primary tumor must be ≥ 12 cm from the anal verge by rigid proctoscopy
* Stage III tumor must have been completely resected within the past 56 days

  * Must have documented en bloc resection in patients with tumor adherence to adjacent structures
  * Tumor-related obstructions and colonic perforation are allowed
  * Tumor samples must be available
* At least 1 pathologically confirmed positive lymph node

  * No evidence of residual involved lymph node disease
* Synchronous primary colon cancer allowed
* No distant metastatic disease
* Performance status - Eastern Cooperative Oncology Group (ECOG) 0-2
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Creatinine ≤ 1.5 times ULN
* No uncontrolled high blood pressure
* No unstable angina
* No symptomatic congestive heart failure
* No myocardial infarction with the past 6 months
* No New York Heart Association class III or IV heart disease
* No symptomatic pulmonary fibrosis
* No symptomatic interstitial pneumonitis
* No prior allergic reaction (known sensitivity) to chimerized or murine monoclonal antibody therapy
* No known allergy to platinum compounds
* No documented presence of human anti-mouse antibodies (HAMA)
* No active uncontrolled bacterial, viral, or systemic fungal infection
* HIV negative
* No clinically defined AIDS
* Not pregnant or nursing
* Negative pregnancy test
* No men or women of childbearing potential who are unwilling to employ adequate contraception
* No inadequately treated gastrointestinal bleeding
* No ≥ grade 2 pre-existing peripheral sensory or motor neuropathy
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or lobular carcinoma in situ in 1 breast
* No other concurrent medical condition that would preclude study participation
* No concurrent biologic therapy
* No prior chemotherapy for colon cancer
* No other concurrent chemotherapy
* No prior radiotherapy for colon cancer
* No concurrent targeted agents
* No prior agents directed against epidermal growth factor-receptor
* No other concurrent anticancer therapy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3397 (Actual)
Dates: Start 2004-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Alberts, MD, Principal Investigator — North Central Cancer Treatment Group
Locations (894):
- United States (858):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Clearview Cancer Institute, Huntsville, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Providence Hospital, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Thunderbird Medical Center, Glendale, Arizona
  - Banner Desert Medical Center, Mesa, Arizona
  - Banner Baywood Medical Center, Mesa, Arizona
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - Western Regional CCOP, Phoenix, Arizona
  - Phoenix Indian Medical Center, Phoenix, Arizona
  - Scottsdale Healthcare, Scottsdale, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Highlands Oncology Group-Bentonville, Bentonville, Arkansas
  - Saint Edward Mercy Medical Center, Fort Smith, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veteran's Administration Medical Center, Little Rock, Arkansas
  - Alta Bates Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center, Burbank, California
  - Mills - Peninsula Hospitals, Burlingame, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - City of Hope, Duarte, California
  - Northbay Cancer Center, Fairfield, California
  - Kaiser Permanente, Fremont, Fremont, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - California Cancer Center - North Fresno, Fresno, California
  - Cancer Care Associates, Fresno, California
  - California Cancer Care - Greenbrae, Greenbrae, California
  - Sutter Health Western Division Cancer Research Group, Greenbrae, California
  - Kaiser Permanente, Hayward, Hayward, California
  - Saint Rose Hospital, Hayward, California
  - Loma Linda University Medical Center, Loma Linda, California
  - University of Southern California, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Memorial Medical Center, Modesto, California
  - Community Hospital of Monterey Peninsula, Monterey, California
  - El Camino Hospital, Mountain View, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Breast Surgeons Inc, Oakland, California
  - Bay Area Tumor Institution CCOP, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Saint Joseph Hospital, Orange, California
  - Desert Regional Medical Center, Palm Springs, California
  - Palo Alto Medical Foundation Heath Care, Palo Alto, California
  - Valley Care Health System - Pleasanton, Pleasanton, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Shasta Regional Medical Center, Redding, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter General Hospital, Sacramento, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Kaiser Permanente, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - University of California San Diego - Veterans Administration, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - University of California San Francisco Medical Center-Mount Zion, San Francisco, California
  - California Pacific Medical Center, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Santa Rosa Memorial Hospital, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Tahoe Forest Cancer Center, Truckee, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Memorial Hospital Colorado Springs, Colorado Springs, Colorado
  - Saint Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Exempla Saint Joseph Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program CCOP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Danbury Hospital, Danbury, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Manchester Memorial Hospital, Manchester, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Stamford Hospital, Stamford, Connecticut
  - Bayhealth Medical Center at Kent General, Dover, Delaware
  - Beebe Medical Center, Lewes, Delaware
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Lombardi Comprehensive Cancer Center at Georgetown University, Washington D.C., District of Columbia
  - Howard University Hospital, Washington D.C., District of Columbia
  - Halifax Medical Center-Centers for Oncology, Daytona Beach, Florida
  - North Broward Medical Center, Deerfield Beach, Florida
  - Broward General Medical Center, Fort Lauderdale, Florida
  - University of Florida, Gainesville, Florida
  - Edna Williams Cancer Center at the Baptist Cancer Institute, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - The Watson Clinic, Lakeland, Florida
  - Cancer Centers of Central Florida PA, Leesburg, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Integrated Community Oncology Network - Orange Park Cancer Center, Orange Park, Florida
  - Florida Hospital, Orlando, Florida
  - M D Anderson Cancer Center- Orlando, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Sacred Heart Medical Oncology Group - Davis Highway, Pensacola, Florida
  - Montgomery and Associates MD PA, Saint Augustine, Florida
  - Florida Cancer Specialists - Sarasota Downtown, Sarasota, Florida
  - Martin Memorial Cancer Center, Stuart, Florida
  - Martin Memorial Medical Center - North, Stuart, Florida
  - Martin Memorial Hospital - South, Stuart, Florida
  - Palm Beach Cancer Institute-Main Office, West Palm Beach, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Atlanta Regional CCOP, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - Augusta Oncology Associates PC, Augusta, Georgia
  - Well Star Cobb Hospital, Austell, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Veterans Administration Medical Center, Decatur, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Saint Joseph's-Candler Health System, Savannah, Georgia
  - South Georgia Medical Center, Valdosta, Georgia
  - Oncare Hawaii Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii, Honolulu, Hawaii
  - Hawaii Medical Center East, Honolulu, Hawaii
  - Oncare Hawaii Inc-Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute of Maui, Wailuku, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Saint Anthony's Health, Alton, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Mercy Hospital and Medical Center, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - Resurrection Healthcare, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Illinois Masonic Medical Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Saint Anthony Memorial Hospital, Effingham, Illinois
  - Sherman Hospital, Elgin, Illinois
  - Cancer Institute at Alexian Brothers, Elk Grove Village, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Evanston CCOP-NorthShore University HealthSystem, Evanston, Illinois
  - Saint Francis Hospital, Evanston, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Intercommunity Cancer Center, Galesburg, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Midwest Center for Hematology Oncology, Joliet, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Provena Saint Mary's Hospital, Kankakee, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - La Grange Memorial Hospital, La Grange, Illinois
  - Deerpath Medical Associates, Lake Forest, Illinois
  - North Shore Hematology Oncology, Libertyville, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Sharis, Christine M MD (UIA Investigator), Moline, Illinois
  - Stoffel, Thomas J MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Vigliotti, Antonio, P.G. M.D. (UIA Investigator), Moline, Illinois
  - Good Samaritan Regional Medical Center, Mount Vernon, Illinois
  - Hematology Oncology Consultants Limited, Naperville, Illinois
  - Edward Hospital, Naperville, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland PC, Niles, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois Oncology Research Association CCOP, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - West Suburban Cancer Center, River Forest, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - Sarah Culbertson Memorial Hospital, Rushville, Illinois
  - Edward H Kaplan MD and Associates, Skokie, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Midwest Cancer Research Group Incorporated, Skokie, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Valley Cancer Center, Spring Valley, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Clinic-Urbana Main, Urbana, Illinois
  - Carle Foundation dba Carle Cancer Center, Urbana, Illinois
  - Saint Francis Hospital and Health Centers, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc - State Boulevard, Fort Wayne, Indiana
  - Indiana University Medical Center, Indianapolis, Indiana
  - Richard L. Roudebush Veterans Affairs Medical Center, Indianapolis, Indiana
  - Wishard Hospital, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Services, Indianapolis, Indiana
  - Howard Regional Healthcare System, Kokomo, Indiana
  - Laporte Hospital, La Porte, Indiana
  - Clarian Arnett Cancer Care, Lafayette, Indiana
  - Premier Oncology Hematology Associates, Merrillville, Indiana
  - Saint Anthony Memorial Health Center, Michigan City, Indiana
  - Ball Memorial Hospital, Muncie, Indiana
  - The Community Hospital, Munster, Indiana
  - Reid Hospital and Health Care Services, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Saint Joseph's Medical Center, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - McFarland Clinic, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - Hematology Oncology Associates-Quad Cities, Bettendorf, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Iowa Blood and Cancer Care PLC, Cedar Rapids, Iowa
  - Saint Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Association, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Genesis Medical Center - West Campus, Davenport, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa Oncology Research Association CCOP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Finley Hospital, Dubuque, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Community Memorial Hospital, Missouri Valley, Iowa
  - Burgess Memorial Hospital, Onawa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Siouxland Hematology - Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Covenant Medical Center, Waterloo, Iowa
  - Memorial Hospital of Arkansas City, Arkansas City, Kansas
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Providence Medical Center, Kansas City, Kansas
  - University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Olathe Medical Center, Olathe, Kansas
  - Cancer Center of Kansas - Ottawa, Ottawa, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Radiation Oncology Practice Corporation Southwest, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Mount Carmel Regional Cancer Center, Pittsburg, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Stormont-Vail Regional Health Center, Topeka, Kansas
  - Saint Francis Hospital and Medical Center - Topeka, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita CCOP, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Our Lady Bellefonte Hospital, Ashland, Kentucky
  - Central Baptist Hospital, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Merle Mahr Cancer Center, Madisonville, Kentucky
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Clinic Foundation-Baton Rouge, Baton Rouge, Louisiana
  - DeSoto Regional Health System, Mansfield, Louisiana
  - Metairie Oncologists, Metairie, Louisiana
  - Louisiana State University Sciences Center- Monroe, Monroe, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Medical Center of Louisiana, New Orleans, Louisiana
  - Ochsner Clinic CCOP, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Highland Clinic, Shreveport, Louisiana
  - Louisiana State University, Shreveport, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - The Union Memorial Hospital, Baltimore, Maryland
  - Franklin Square Hospital Center, Baltimore, Maryland
  - Good Samaritan Hospital of Maryland, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Washington County Hospital, Hagerstown, Maryland
  - Associates in Oncology Hematology PC -Kensington, Kensington, Maryland
  - Associates In Oncology Hematology PC-Rockville, Rockville, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Caritas Saint Elizabeth's Medical Center, Brighton, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Franklin Medical Center, Greenfield, Massachusetts
  - Holyoke Medical Center, Holyoke, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Lawrence Memorial, Medford, Massachusetts
  - Holy Family Hospital, Methuen, Massachusetts
  - Metrowest Medical Center Incorporated, Natick, Massachusetts
  - Norwood Hospital, Norwood, Massachusetts
  - North Shore Medical Center Cancer Center, Peabody, Massachusetts
  - Berkshire Hematology Oncology PC, Pittsfield, Massachusetts
  - Commonwealth Hematology Oncology PC-Quincy, Quincy, Massachusetts
  - South Shore Hospital, South Weymouth, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Morton Hospital and Medical Center, Taunton, Massachusetts
  - Noble Hospital, Westfield, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium Community Clinical Oncology Program, Ann Arbor, Michigan
  - Battle Creek Health System, Battle Creek, Michigan
  - Bay Regional Medical Center, Bay City, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Hospital, Dearborn, Michigan
  - Wayne State University, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Michigan State University - Breslin Cancer Center, East Lansing, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center, Flint, Michigan
  - McLaren Regional Medical Center, Flint, Michigan
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Saint Mary's Health Care, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Spectrum Health-Blodgett Campus, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - Ingham Regional Medical Center, Lansing, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Lapeer Regional Hospital, Lapeer, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mid-Michigan Medical Center - Midland, Midland, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Mercy Health Partners-Hackley Campus, Muskegon, Michigan
  - Mercy Health Partners-Mercy Campus, Muskegon, Michigan
  - Northern Michigan Regional Hospital, Petoskey, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Providence Hospital, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Harris, John Gilbert MD (UIA Investigator), Alexandria, Minnesota
  - Medini, Eitan MD (UIA Investigator), Alexandria, Minnesota
  - Merit Care Clinic Bemidji, Bemidji, Minnesota
  - Brainerd Medical Center Inc, Brainerd, Minnesota
  - Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic CCOP, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Saint Mary's Medical Center, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Etzell, Paul S MD (UIA Investigator), Fergus Falls, Minnesota
  - Swenson, Wade II, MD (UIA Investigator), Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - Immanuel-Saint Joseph Hospital-Mayo Health System, Mankato, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Minneapolis Veterans Medical Center, Minneapolis, Minnesota
  - Chippewa County - Montevideo Hospital, Montevideo, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro-Minnesota CCOP, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Joseph's Hospital - Healtheast, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Adult and Pediatric Urology PLLP, Sartell, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - Veterans Affairs Medical Center, Jackson, Mississippi
  - Keesler Medical Center, Keesler Air Force Base, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Missouri Cancer Associates, Columbia, Missouri
  - Independence Regional Health Center, Independence, Missouri
  - Freeman Health System, Joplin, Missouri
  - Saint John's Regional Medical Center, Joplin, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Radiation Oncology Practice Corporation South, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - Liberty Radiation Oncology Clinic, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Radiation Oncology Practice Corporation - North, Kansas City, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Missouri Cancer Care PC - Saint Charles, Saint Charles, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Ozark Health Ventures LLC dba Cancer Research for The Ozarks Springfield, Springfield, Missouri
  - Saint John's Hospital, Springfield, Missouri
  - Cox Medical Center, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute, St Louis, Missouri
  - Saint Louis University Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Saint Anthony's Medical Center, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Christian Hospital Northeast - Northwest, St Louis, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - Saint John's Mercy Medical Center, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Hematology-Oncology Centers of the Northern Rockies PC, Billings, Montana
  - Montana Cancer Consortium CCOP, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Billings Clinic, Billings, Montana
  - Deaconess Medical Center, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Internal Medicine of Bozeman, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Eastern Montana Cancer Center, Miles City, Montana
  - Community Medical Hospital, Missoula, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Fremont Area Medical Center, Fremont, Nebraska
  - Saint Francis Medical Center, Grand Island, Nebraska
  - Good Samaritan Hospital, Kearney, Nebraska
  - Bryan LGH Medical Center West, Lincoln, Nebraska
  - Bryan LGH Medical Center East, Lincoln, Nebraska
  - Lincoln Medical Education Foundation Cancer Resource Center, Lincoln, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Great Plains Regional Medical Center, North Platte, Nebraska
  - Missouri Valley Cancer Consortium CCOP, Omaha, Nebraska
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Nevada Cancer Institute, Las Vegas, Nevada
  - New Hampshire Oncology-Hematology PA, Concord, New Hampshire
  - Columbia Parkland Medical Center, Derry, New Hampshire
  - Exeter Hospital, Exeter, New Hampshire
  - New Hampshire Oncology Hematology Associates, Hooksett, New Hampshire
  - Cheshire Medical Center-Dartmouth-Hitchcock Keene, Keene, New Hampshire
  - LRGHealthcare-Lakes Region General Hospital, Laconia, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Elliot Hospital, Manchester, New Hampshire
  - Portsmouth Regional Hospital, Portsmouth, New Hampshire
  - Ocean Medical Center, Brick, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Hunterdon Medical Center, Flemington, New Jersey
  - CentraState Medical Center, Freehold, New Jersey
  - Cancer Institute of New Jersey At Hamilton, Hamilton, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Mountainside Hospital, Montclair, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital of Burlington County, Mount Holly, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Warren Hospital, Phillipsburg, New Jersey
  - Booker Cancer Center at Riverview Medical Center, Red Bank, New Jersey
  - Somerset Medical Center, Somerville, New Jersey
  - Sparta Cancer Treatment Center, Sparta, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - South Jersey Healthcare, Vineland, New Jersey
  - Virtua West Jersey Hospital Voorhees, Voorhees Township, New Jersey
  - University of New Mexico at Lovelace Medical Center, Albuquerque, New Mexico
  - Hematology Oncology Associates, Albuquerque, New Mexico
  - University of New Mexico, Albuquerque, New Mexico
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico
  - Long Island College Hospital, Brooklyn, New York
  - Veterans Affairs Western New York Health Care System-Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Hematology Oncology Associates of Central New York, East Syracuse, New York
  - Adirondack Cancer Center, Glens Falls, New York
  - Catskill Regional Medical Center, Harris, New York
  - Orange Regional Medical Center, Middletown, New York
  - Winthrop University Hospital, Mineola, New York
  - Beth Israel Medical Center, New York, New York
  - New York University Langone Medical Center, New York, New York
  - Saint Luke's Roosevelt Hospital Center - Saint Luke's Division, New York, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Nyack Hospital, Nyack, New York
  - Highland Hospital, Rochester, New York
  - Interlakes Foundation Inc-Rochester, Rochester, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - The North Division of Montefiore Medical Center, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Faxton-Saint Luke's Healthcare, Utica, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - Mission Hospitals Inc, Asheville, North Carolina
  - Alamance Regional Medical Center, Burlington, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Gaston Memorial Hospital, Gastonia, North Carolina
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Marion L Shepard Cancer Center, Washington, North Carolina
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Health Systems, Bismarck, North Dakota
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Veterans Administration Medical Center, Fargo, North Dakota
  - Innovis Health South University, Fargo, North Dakota
  - Meritcare Hospital, Fargo, North Dakota
  - MeritCare Medical Group, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Akron City Hospital, Akron, Ohio
  - Akron General Medical Center, Akron, Ohio
  - Summa Barberton Hospital, Barberton, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - The Boardman Cancer Center, Boardman, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Mercy Medical Center, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus CCOP, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Veteran Affairs Medical Center, Dayton, Ohio
  - Dayton CCOP, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Cole, Sharon, K. M.D. (UIA Investigator), Kenton, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Mansfield General Hospital-MedCentral Health System, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - Saint Luke's Hospital, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Bayview Oncology Associates, Oregon, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Cancer Care Center, Incorporated, Salem, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Community Hospital Springfield, Springfield, Ohio
  - Flower Memorial Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Cancer Center at Saint Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Joseph Cancer Center, Warren, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Cleveland Clinic Wooster Specialty Center, Wooster, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Saint Elizabeth Hospital Medical Center, Youngstown, Ohio
  - Genesis HealthCare System, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research - Lawton, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Cancer Care Associates, Oklahoma City, Oklahoma
  - Natalie W Bryant Cancer Center, Tulsa, Oklahoma
  - Bay Area Hospital, Coos Bay, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - Columbia River Oncology Program, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Northwest Cancer Specialists-Rose Quarter Cancer Center, Portland, Oregon
  - Kaiser Permanente, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Salem Hospital, Salem, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Saint Luke's Hospital, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Marion Community Hospital, Carbondale, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Easton Hospital, Easton, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - PinnacleHealth Regional Cancer Center at Polyclinic Hospital, Harrisburg, Pennsylvania
  - Geisinger South Wilkes Barre-Hazelton Cancer Center, Hazleton, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Central PA Hematology-Medical Oncology Associates PC, Lemoyne, Pennsylvania
  - Riddle Hospital, Media, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Abramson Cancer Center of The University of Pennsylvania, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Aria Health-Torresdale Campus, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Pottstown Memorial Medical Center, Pottstown, Pennsylvania
  - Saint Joseph Medical Center, Reading, Pennsylvania
  - Guthrie Clinic - Sayre, Sayre, Pennsylvania
  - Mercy Hospital, Scranton, Pennsylvania
  - Hematology and Oncology Associates of North East Pennsylvania, Scranton, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Moses Taylor Hospital, Scranton, Pennsylvania
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Associates In Hematology Oncology PC-Upland, Upland, Pennsylvania
  - Jennersville Regional Hospital, West Grove, Pennsylvania
  - Reading Hospital and Medical Center, West Reading, Pennsylvania
  - Geisinger Wyoming Valley, Wilkes-Barre, Pennsylvania
  - Lankenau Hospital, Wynnewood, Pennsylvania
  - Mainline Health CCOP, Wynnewood, Pennsylvania
  - Hematology and Oncology Associates of Rhode Island Inc, Cranston, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - Kent County Hospital, Warwick, Rhode Island
  - AnMed Health Hospital, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville CCOP, Greenville, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Upstate Carolina CCOP, Spartanburg, South Carolina
  - Conklin Regional Cancer Center, Aberdeen, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center-Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Sanford University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - Tennessee Oncology PLLC- Centennial Medical Center, Nashville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Texas Health Presbyterian Hospital Dallas, Dallas, Texas
  - The Center for Integrative Cancer Medicine, El Paso, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Methodist Hospital, Houston, Texas
  - Saint Luke's Episcopal Hospital, Houston, Texas
  - Veterans Administration Medical Center, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Doctor's Hospital of Laredo, Laredo, Texas
  - Audie L Murphy Veterans Affairs Hospital, San Antonio, Texas
  - University of Texas Health Science Center, San Antonio, Texas
  - Cancer Therapy and Research Center at The UT Health Science Center at San Antonio, San Antonio, Texas
  - South Texas Oncology and Hematology PA, San Antonio, Texas
  - University Hospital, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Southwestern Oncology Research Department, Bennington, Vermont
  - University of Vermont, Burlington, Vermont
  - Danville Regional Medical Center, Danville, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Riverside Middle Peninsula Cancer Center, Gloucester, Virginia
  - Lynchburg Hematology-Oncology Clinic, Lynchburg, Virginia
  - Peninsula Cancer Institute-Newport News, Newport News, Virginia
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - Peninsula Cancer Institute, Williamsburg, Virginia
  - Auburn Regional Medical Center, Auburn, Washington
  - Saint Joseph Hospital, Bellingham, Washington
  - Harrison Bremerton Hematology and Oncology, Bremerton, Washington
  - Providence Centralia Hospital, Centralia, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Columbia Basin Hematology and Oncology PLLC, Kennewick, Washington
  - Evergreen Hospital Medical Center, Kirkland, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - Capital Medical Center, Olympia, Washington
  - Olympic Medical Center, Port Angeles, Washington
  - Good Samaritan Community Hospital, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - Virginia Mason CCOP, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Puget Sound Oncology Consortium, Seattle, Washington
  - Group Health Cooperative, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - The Polyclinic, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Sacred Heart Medical Center, Spokane, Washington
  - Holy Family Hospital, Spokane, Washington
  - Allenmore Hospital, Tacoma, Washington
  - Northwest CCOP, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Tacoma General Hospital, Tacoma, Washington
  - Multicare Health System, Tacoma, Washington
  - Saint Clare Hospital, Tacoma, Washington
  - Southwest Washington Medical Center, Vancouver, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - West Virginia University, Morgantown, West Virginia
  - Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - Princeton Community Hospital, Princeton, West Virginia
  - Wheeling Hospital, Wheeling, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Sacred Heart Hospital, Eau Claire, Wisconsin
  - Midelfort Clinic-Clairemont Campus, Eau Claire, Wisconsin
  - Mayo Clinic Health System Eau Claire Hospital - Luther Campus, Eau Claire, Wisconsin
  - Central Wisconsin Cancer Program, Fond du Lac, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercy Health System, Janesville, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Franciscan Skemp Healthcare, La Crosse, Wisconsin
  - UW Health Oncology - 1 South Park, Madison, Wisconsin
  - Dean Hematology and Oncology Clinic, Madison, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Vince Lombardi Cancer Clinic-Marinette, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Oconomowoc Memorial Hospital-ProHealth Care Inc, Oconomowoc, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Marshfield Clinic at James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (31):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Lions Gate Hospital, North Vancouver, British Columbia
  - BCCA-Fraser Valley Cancer Centre, Surrey, British Columbia
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - The Moncton Hospital, Moncton, New Brunswick
  - Atlantic Health Sciences Corporation-Saint John Regional Hospital, Saint John, New Brunswick
  - The Royal Victoria Hospital, Barrie, Ontario
  - Cambridge Memorial Hospital, Cambridge, Ontario
  - Regional Cancer Program of The Hopital Regional de Sudbury Regional Hopital, Greater Sudbury, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Grand River Regional Cancer Centre at Grand River Hospital, Kitchener, Ontario
  - London Regional Cancer Program, London, Ontario
  - Credit Valley Hospital, Mississauga, Ontario
  - Ottawa Health Research Institute-General Division, Ottawa, Ontario
  - Algoma District Cancer Program Sault Area Hospital, Sault Ste. Marie, Ontario
  - Niagara Health System-Saint Catharines General, St. Catharines, Ontario
  - Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Saint Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Trillium Health Centre-West Toronto, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - PEI Cancer Treatment Centre-Queen Elizabeth Hospital, Charlottetown, Prince Edward Island
  - McGill University Department of Oncology, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Puerto Rico (5):
  - Andres Grillasca Hospital, Ponce
  - Hato Rey Hematology Oncology Group, San Juan
  - I Gonzales Martinez-Oncologic Hospital, San Juan
  - San Juan Veterans Affairs Medical Center, San Juan
  - San Juan City Hospital, San Juan

REFERENCES:
- [Derived] Gallois C, Shi Q, Meyers JP, Iveson T, Alberts SR, de Gramont A, Sobrero AF, Haller DG, Oki E, Shields AF, Goldberg RM, Kerr R, Lonardi S, Yothers G, Kelly C, Boukovinas I, Labianca R, Sinicrope FA, Souglakos I, Yoshino T, Meyerhardt JA, Andre T, Papamichael D, Taieb J. Prognostic Impact of Early Treatment and Oxaliplatin Discontinuation in Patients With Stage III Colon Cancer: An ACCENT/IDEA Pooled Analysis of 11 Adjuvant Trials. J Clin Oncol. 2023 Feb 1;41(4):803-815. doi: 10.1200/JCO.21.02726. Epub 2022 Oct 28. PMID 36306483
- [Derived] Saberzadeh-Ardestani B, Foster NR, Lee HE, Shi Q, Alberts SR, Smyrk TC, Sinicrope FA. Association of tumor-infiltrating lymphocytes with survival depends on primary tumor sidedness in stage III colon cancers (NCCTG N0147) [Alliance]. Ann Oncol. 2022 Nov;33(11):1159-1167. doi: 10.1016/j.annonc.2022.07.1942. Epub 2022 Aug 10. PMID 35963480
- [Derived] Azizi Z, Zheng C, Mosquera L, Pilote L, El Emam K; GOING-FWD Collaborators. Can synthetic data be a proxy for real clinical trial data? A validation study. BMJ Open. 2021 Apr 16;11(4):e043497. doi: 10.1136/bmjopen-2020-043497. PMID 33863713
- [Derived] Cohen R, Taieb J, Fiskum J, Yothers G, Goldberg R, Yoshino T, Alberts S, Allegra C, de Gramont A, Seitz JF, O'Connell M, Haller D, Wolmark N, Erlichman C, Zaniboni A, Lonardi S, Kerr R, Grothey A, Sinicrope FA, Andre T, Shi Q. Microsatellite Instability in Patients With Stage III Colon Cancer Receiving Fluoropyrimidine With or Without Oxaliplatin: An ACCENT Pooled Analysis of 12 Adjuvant Trials. J Clin Oncol. 2021 Feb 20;39(6):642-651. doi: 10.1200/JCO.20.01600. Epub 2020 Dec 23. PMID 33356421
- [Derived] Labadie JD, Hua X, Harrison TA, Banbury BL, Huyghe JR, Sun W, Shi Q, Yothers G, Alberts SR, Sinicrope FA, Goldberg RM, George TJ, Penney KL, Phipps AI, Cohen SA, Peters U, Chan AT, Newcomb PA. Genetic Predictors of Severe Skin Toxicity in Patients with Stage III Colon Cancer Treated with Cetuximab: NCCTG N0147 (Alliance). Cancer Epidemiol Biomarkers Prev. 2021 Feb;30(2):404-411. doi: 10.1158/1055-9965.EPI-20-1274. Epub 2020 Nov 17. PMID 33203692
- [Derived] Lee H, Sha D, Foster NR, Shi Q, Alberts SR, Smyrk TC, Sinicrope FA. Analysis of tumor microenvironmental features to refine prognosis by T, N risk group in patients with stage III colon cancer (NCCTG N0147) (Alliance). Ann Oncol. 2020 Apr;31(4):487-494. doi: 10.1016/j.annonc.2020.01.011. Epub 2020 Jan 25. PMID 32165096
- [Derived] Penney KL, Banbury BL, Bien S, Harrison TA, Hua X, Phipps AI, Sun W, Song M, Joshi AD, Alberts SR, Allegra CJ, Atkins J, Colangelo LH, George TJ, Goldberg RM, Lucas PC, Nair SG, Shi Q, Sinicrope FA, Wolmark N, Yothers G, Peters U, Newcomb PA, Chan AT. Genetic Variant Associated With Survival of Patients With Stage II-III Colon Cancer. Clin Gastroenterol Hepatol. 2020 Nov;18(12):2717-2723.e3. doi: 10.1016/j.cgh.2019.11.046. Epub 2019 Dec 4. PMID 31811950
- [Derived] Taieb J, Shi Q, Pederson L, Alberts S, Wolmark N, Van Cutsem E, de Gramont A, Kerr R, Grothey A, Lonardi S, Yoshino T, Yothers G, Sinicrope FA, Zaanan A, Andre T. Prognosis of microsatellite instability and/or mismatch repair deficiency stage III colon cancer patients after disease recurrence following adjuvant treatment: results of an ACCENT pooled analysis of seven studies. Ann Oncol. 2019 Sep 1;30(9):1466-1471. doi: 10.1093/annonc/mdz208. PMID 31268130
- [Derived] Zaanan A, Shi Q, Taieb J, Alberts SR, Meyers JP, Smyrk TC, Julie C, Zawadi A, Tabernero J, Mini E, Goldberg RM, Folprecht G, Van Laethem JL, Le Malicot K, Sargent DJ, Laurent-Puig P, Sinicrope FA. Role of Deficient DNA Mismatch Repair Status in Patients With Stage III Colon Cancer Treated With FOLFOX Adjuvant Chemotherapy: A Pooled Analysis From 2 Randomized Clinical Trials. JAMA Oncol. 2018 Mar 1;4(3):379-383. doi: 10.1001/jamaoncol.2017.2899. PMID 28983557
- [Derived] Sinicrope FA, Shi Q, Allegra CJ, Smyrk TC, Thibodeau SN, Goldberg RM, Meyers JP, Pogue-Geile KL, Yothers G, Sargent DJ, Alberts SR. Association of DNA Mismatch Repair and Mutations in BRAF and KRAS With Survival After Recurrence in Stage III Colon Cancers : A Secondary Analysis of 2 Randomized Clinical Trials. JAMA Oncol. 2017 Apr 1;3(4):472-480. doi: 10.1001/jamaoncol.2016.5469. PMID 28006055
- [Derived] Sticca RP, Alberts SR, Mahoney MR, Sargent DJ, Finstuen LM, Nelson GD, Husted TM, Franko J, Goldman CD, Pockaj BA. Current use and surgical efficacy of laparoscopic colectomy in colon cancer. J Am Coll Surg. 2013 Jul;217(1):56-62; discussion 62-3. doi: 10.1016/j.jamcollsurg.2013.02.023. Epub 2013 Apr 24. PMID 23623224
- [Derived] Alberts SR, Sargent DJ, Nair S, Mahoney MR, Mooney M, Thibodeau SN, Smyrk TC, Sinicrope FA, Chan E, Gill S, Kahlenberg MS, Shields AF, Quesenberry JT, Webb TA, Farr GH Jr, Pockaj BA, Grothey A, Goldberg RM. Effect of oxaliplatin, fluorouracil, and leucovorin with or without cetuximab on survival among patients with resected stage III colon cancer: a randomized trial. JAMA. 2012 Apr 4;307(13):1383-93. doi: 10.1001/jama.2012.385. PMID 22474202
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm E (Combination Chemotherapy, Monoclonal Antibody): Patients received cetuximab as in arm D and irinotecan, leucovorin calcium, and fluorouracil as in arm B. Treatment repeated every 14 days for up to 12 courses in the absence of unacceptable toxicity or recurrent disease.
  irinotecan hydrochloride: Given IV
  leucovorin calcium: Given IV
  fluorouracil: Given I
  cetuximab: Given IV
- Arm G (Locally Directed Therapy): Patients determined to have mutated Kirsten rat sarcoma (KRAS) (or KRAS not evaluable) were assigned to an event monitoring arm in which adjuvant therapy was determined and assigned by the treating oncologist. The determination of the type of therapy, duration of treatment, and dose modification was the responsibility of the treating oncologists.
  Locally Directed Therapy: Patients determined to have mutated KRAS (or KRAS not evaluable) were assigned to an event monitoring arm in which adjuvant therapy was determined and assigned by the treating oncologist. The determination of the type of therapy, duration of treatment, and dose modification was the responsibility of the treating oncologists.
Period: Overall Study
Arm/Group | Arm A (Combination Chemotherapy) | Arm B (Combination Chemotherapy) | Arm C (Combination Chemotherapy) | Arm D (Combination Chemotherapy, Monoclonal Antibody) | Arm E (Combination Chemotherapy, Monoclonal Antibody) | Arm F (Combination Chemotherapy, Monoclonal Antibody) | Arm G (Locally Directed Therapy)
Started | 1402 | 111 | 111 | 1350 | 45 | 46 | 332
Completed | 1081 | 84 | 84 | 906 | 30 | 26 | 332
Not Completed | 321 | 27 | 27 | 444 | 15 | 20 | 0
Not completed — Withdrawal by Subject | 111 | 10 | 12 | 163 | 7 | 8 | 0
Not completed — Adverse Event | 130 | 8 | 8 | 184 | 7 | 8 | 0
Not completed — Recurrence | 21 | 0 | 1 | 15 | 0 | 2 | 0
Not completed — Alternate Treatment | 6 | 1 | 0 | 3 | 0 | 0 | 0
Not completed — Other Medical Problems | 6 | 1 | 0 | 7 | 0 | 0 | 0
Not completed — Death | 4 | 0 | 1 | 15 | 0 | 0 | 0
Not completed — Cytogenetic resistance | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Other | 43 | 7 | 5 | 55 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm G (Locally Directed Therapy): Patients determined to have mutated KRAS (or KRAS not evaluable) were assigned to an event monitoring arm in which adjuvant therapy was determined and assigned by the treating oncologist. The determination of the type of therapy, duration of treatment, and dose modification was the responsibility of the treating oncologists.
  Locally Directed Therapy: Patients determined to have mutated KRAS (or KRAS not evaluable) were assigned to an event monitoring arm in which adjuvant therapy was determined and assigned by the treating oncologist. The determination of the type of therapy, duration of treatment, and dose modification was the responsibility of the treating oncologists.
- Total: Total of all reporting groups
Arm/Group | Arm A (Combination Chemotherapy) | Arm B (Combination Chemotherapy) | Arm C (Combination Chemotherapy) | Arm D (Combination Chemotherapy, Monoclonal Antibody) | Arm E (Combination Chemotherapy, Monoclonal Antibody) | Arm F (Combination Chemotherapy, Monoclonal Antibody) | Arm G (Locally Directed Therapy) | Total
Number analyzed (Participants) | 1402 | 111 | 111 | 1350 | 45 | 46 | 332 | 3397
Age, Continuous [Median (Full Range); unit: years] | 58 [19 to 85] | 57 [25 to 82] | 60 [24 to 82] | 58 [22 to 86] | 59 [30 to 82] | 60.5 [30 to 81] | 56 [22 to 84] | 58 [19 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 662 | 53 | 50 | 647 | 20 | 21 | 160 | 1613
  Male | 740 | 58 | 61 | 703 | 25 | 25 | 172 | 1784
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 64 | 5 | 3 | 62 | 4 | 2 | 18 | 158
  Not Hispanic or Latino | 1107 | 103 | 103 | 1060 | 38 | 41 | 225 | 2677
  Unknown or Not Reported | 231 | 3 | 5 | 228 | 3 | 3 | 89 | 562
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 1 | 1 | 7 | 0 | 0 | 1 | 16
  Asian | 66 | 4 | 2 | 62 | 3 | 0 | 12 | 149
  Native Hawaiian or Other Pacific Islander | 8 | 0 | 1 | 7 | 0 | 0 | 0 | 16
  Black or African American | 94 | 6 | 7 | 96 | 5 | 2 | 29 | 239
  White | 1202 | 98 | 100 | 1154 | 37 | 43 | 275 | 2909
  More than one race | 3 | 2 | 0 | 3 | 0 | 0 | 1 | 9
  Unknown or Not Reported | 23 | 0 | 0 | 21 | 0 | 1 | 14 | 59
Region of Enrollment [Number; unit: participants]
  United States | 1258 | 109 | 109 | 1224 | 44 | 46 | 303 | 3093
  Canada | 138 | 2 | 2 | 124 | 1 | 0 | 28 | 295
  Jamaica | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Puerto Rico | 5 | 0 | 0 | 2 | 0 | 0 | 1 | 8
Positive Nodes [Number; unit: participants] — Number of positive nodes
  participants
    1-3 | 816 | 71 | 70 | 790 | 29 | 28 | 203 | 2007
    4+ | 586 | 40 | 41 | 560 | 16 | 18 | 129 | 1390
Tumor Stage [Number; unit: participants] — T1: Tumor invades submucosa
  T2: Tumor invades muscularis propria
  T3: Tumor invades through the muscularis propria into the subserosa or into non-peritonealized pericolic or perirectal tissues
  T4: (T4a+) Tumor perforates the visceral peritoneum without adherence to or invasion of other organs or structures or (T4b) Tumor is adherent to or directly invades other organs or structures
  participants
    T1 or T2 | 198 | 18 | 14 | 213 | 5 | 5 | 56 | 509
    T3 | 1046 | 78 | 93 | 983 | 35 | 39 | 214 | 2488
    T4 | 158 | 15 | 4 | 153 | 4 | 2 | 62 | 398
    Not Availabe | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Histologic Grade [Number; unit: participants] — High=poorly differentiated or undifferentiated> Low=well or moderately differentiated
  participants
    High | 357 | 25 | 28 | 345 | 10 | 12 | 60 | 837
    Low | 1045 | 86 | 83 | 1005 | 35 | 34 | 272 | 2560
KRAS Status [Number; unit: participants]
  Unknown | 56 | 6 | 6 | 51 | 3 | 4 | 6 | 132
  Mutant | 391 | 33 | 43 | 345 | 15 | 13 | 326 | 1166
  Wildtype | 955 | 72 | 62 | 954 | 27 | 29 | 0 | 2099

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival (Arms A and D: Wild-type KRAS Patients)
Description: The primary endpoint for this study was to compare the disease-free survival (DFS) in patients with stage III colon cancer who are KRAS wild-type randomized to one of two treatment regimens: 1) oxaliplatin, leucovorin calcium, and fluorouracil (Arm A) or 2) oxaliplatin, leucovorin calcium, fluorouracil and cetuximab (Arm D). Participants treated according to Arms B, C, E, and F treatment schedules received treatment which included irinotecan hydrochloride and therefore were not analyzed for this endpoint.
  Disease-free survival is defined as the time from randomization until tumor recurrence or death, whichever is first. Estimated by the method of Kaplan and Meier.
Time Frame: At 3 years
Population: The analysis was performed using intention to treat principles. All patients that were wild-type KRAS and received randomized treatment according to the Arm A or Arm D intervention schedule were evaluated for this endpoint. Any patient receiving irinotecan was not included in the evaluation of this endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Wild-type KRAS Arm A: Patients from Arm A (and a few patients from Arm C that did not receive irinotecan) that are wild-type KRAS and concurrently randomized with Arm D patients.
- Wild-type KRAS Arm D: Patients from Arm D (and a few patients from Arm F that did not receive irinotecan) that are wild-type KRAS and concurrently randomized with Arm A patients.
Arm/Group | Wild-type KRAS Arm A | Wild-type KRAS Arm D
Number analyzed (Participants) | 909 | 954
percentage of participants | 74.6 [71.1 to 78.3] | 71.5 [67.8 to 75.4]

2. Secondary Outcome: Disease-free Survival (Arms A and D: Mutant KRAS Patients)
Description: A secondary endpoint for this study was to investigate the disease-free survival (DFS) in patients with stage III colon cancer who are KRAS mutant (or KRAS-nonevaluable) and randomized to one of two treatment regimens: 1) oxaliplatin, leucovorin calcium, and fluorouracil (Arm A) or 2) oxaliplatin, leucovorin calcium, fluorouracil and cetuximab (Arm D). Participants treated according to Arms B, C, E, and F treatment schedules received treatment which included irinotecan hydrochloride and therefore were not analyzed for this endpoint.
  Disease-free survival is defined as the time from randomization until tumor recurrence or death, whichever is first. Estimated by the method of Kaplan and Meier.
Time Frame: At 3 years
Population: The analysis was performed using intention to treat principles. All patients that were KRAS mutant (or not evaluable for KRAS) and received randomized treatment according to the Arm A or Arm D intervention schedule were evaluated for this endpoint. Any patient receiving irinotecan was not included in the evaluation of this endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Mutant KRAS Arm A: Patients from Arm A (and a few patients from Arm C that did not receive irinotecan) that are mutant KRAS and concurrently randomized with Arm D patients.
- Mutant KRAS Arm D: Patients from Arm D (and a few patients from Arm F that did not receive irinotecan) that are mutant KRAS and concurrently randomized with Arm A patients.
Arm/Group | Mutant KRAS Arm A | Mutant KRAS Arm D
Number analyzed (Participants) | 374 | 343
percentage of participants | 67.1 [61.8 to 72.8] | 65.0 [59.8 to 70.7]

3. Secondary Outcome: Overall Survival as Measured by the 3-year Event-free Rate (Arms A and D: Wild-type KRAS Patients)
Description: Evidence of death from any cause within 3 years counted as events in the time to event- Kaplan Meier analysis of overall survival for patients with stage III colon cancer who are KRAS wild-type randomized to one of two treatment regimens: 1) oxaliplatin, leucovorin calcium, and fluorouracil (Arm A) or 2) oxaliplatin, leucovorin calcium, fluorouracil and cetuximab (Arm D). Participants treated according to Arms B, C, E, and F treatment schedules received treatment which included irinotecan hydrochloride and therefore were not analyzed for this endpoint. The 3-year event free rates (percentage) are reported below for Wild-type KRAS Patients.
Time Frame: Up to 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Wild-type KRAS Arm A | Wild-type KRAS Arm D
Number analyzed (Participants) | 909 | 954
percentage of participants | 87.3 [84.3 to 90.3] | 85.6 [82.7 to 88.7]
Statistical Analysis 1: Comparison: Wild-type KRAS Arm A vs Wild-type KRAS Arm D; Test type: Superiority; p = 0.15, Regression, Cox; HR and p-value reported from a multivariate Cox PH regression model, adjusted for number of nodes, histologic grade, and T stage; Hazard Ratio (HR) = 1.25, 95% CI 2-sided [0.92 to 1.68]

4. Secondary Outcome: Overall Survival as Measured by the 3-year Event-free Rate (Arms A and D: Mutant KRAS Patients)
Description: Evidence of death from any cause within 3 years counted as events in the time to event- Kaplan Meier analysis of overall survival for patients with stage III colon cancer who are KRAS mutant (or KRAS-nonevaluable) and randomized to one of two treatment regimens: 1) oxaliplatin, leucovorin calcium, and fluorouracil (Arm A) or 2) oxaliplatin, leucovorin calcium, fluorouracil and cetuximab (Arm D). Participants treated according to Arms B, C, E, and F treatment schedules received treatment which included irinotecan hydrochloride and therefore were not analyzed for this endpoint. The 3-year event-free rates (percentage) are report below for mutant KRAS patients.
Time Frame: Up to 3 years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mutant KRAS Arm A | Mutant KRAS Arm D
Number analyzed (Participants) | 374 | 343
percentage of participants | 87.9 [84.0 to 91.9] | 82.7 [78.0 to 87.6]
Statistical Analysis 1: Comparison: Mutant KRAS Arm A vs Mutant KRAS Arm D; Test type: Superiority; p = 0.25, Regression, Cox; [statistical method as in outcome 3, analysis 1]; Hazard Ratio (HR) = 1.27, 95% CI 2-sided [0.85 to 1.92]

5. Secondary Outcome: Toxicity, Assessed Using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 (v3) (Arms A and D: Wild-type KRAS Patients)
Description: The maximum grade for each type of toxicity will be recorded for each patient with stage III colon cancer who are KRAS wild-type randomized to one of two treatment regimens: 1) oxaliplatin, leucovorin calcium, and fluorouracil (Arm A) or 2) oxaliplatin, leucovorin calcium, fluorouracil and cetuximab (Arm D). The overall toxicity rates (percentages) for grade 3 or higher adverse events considered at least possibly related to treatment are reported below.
Time Frame: Assessed up to 8 years
Population: All patients that were wild-type KRAS and received randomized treatment according to the Arm A or Arm D intervention schedule and completed the adverse event form at least once were evaluated for this endpoint.
Measure: Number; unit: percentage of patients
Arm/Group | Wild-type KRAS Arm A | Wild-type KRAS Arm D
Number analyzed (Participants) | 894 | 931
percentage of patients | 51.1 | 73.3
Statistical Analysis 1: Comparison: Wild-type KRAS Arm A vs Wild-type KRAS Arm D; Test type: Superiority; p < 0.001, Chi-squared; two-sided chi-squared test

6. Secondary Outcome: Toxicity, Assessed Using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 (v3) (Arms A and D: Mutant KRAS Patients)
Description: The maximum grade for each type of toxicity will be recorded for each patient with stage III colon cancer who are KRAS mutant (or KRAS-nonevaluable) and randomized to one of two treatment regimens: 1) oxaliplatin, leucovorin calcium, and fluorouracil (Arm A) or 2) oxaliplatin, leucovorin calcium, fluorouracil and cetuximab (Arm D). The overall toxicity rates (percentages) for grade 3 or higher adverse events considered at least possibly related to treatment are reported below.
Time Frame: Assessed up to 8 years
Population: All patients that were mutant KRAS and received randomized treatment according to the Arm A or Arm D intervention schedule and completed the adverse event form at least once were evaluated for this endpoint.
Measure: Number; unit: percentage of patients
Arm/Group | Mutant KRAS Arm A | Mutant KRAS Arm D
Number analyzed (Participants) | 367 | 342
percentage of patients | 55.6 | 72.3
Statistical Analysis 1: Comparison: Mutant KRAS Arm A vs Mutant KRAS Arm D; Test type: Superiority; p < 0.001, Chi-squared; Two-sided chi-squared test

ADVERSE EVENTS:
Time Frame: 6 months or during treatment
Description: All patients that received protocol treatment and completed at least one adverse event assessment are included in this analysis. Adverse event data was not collected for Arm G patients.
Groups:
- Arm A (Combination Chemotherapy): Patients receive oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, and fluorouracil IV continuously over 46-48 hours on days 1. Treatment repeats every 14 days for up to 12 courses in the absence of unacceptable toxicity or recurrent disease.
  oxaliplatin: Given IV
  leucovorin calcium: Given IV
  fluorouracil: Given IV
- Arm B (Combination Chemotherapy): Patients receive irinotecan IV over 2 hours on day 1 and leucovorin calcium and fluorouracil as in arm A. Treatment repeats every 14 days for up to 12 courses in the absence of unacceptable toxicity or recurrent disease.
  irinotecan hydrochloride: Given IV
  leucovorin calcium: Given IV
  fluorouracil: Given IV
- Arm C (Combination Chemotherapy): Patients receive the same treatment as in arm A for 6 courses followed by the same treatment as in arm B for 6 courses (total of 12 courses). Treatment continues in the absence of unacceptable toxicity or recurrent disease.
  irinotecan hydrochloride: Given IV
  oxaliplatin: Given IV
  leucovorin calcium: Given IV
  fluorouracil: Given IV
- Arm D (Combination Chemotherapy, Monoclonal Antibody): Patients receive cetuximab IV over 1 hour on days 1 and 8 and oxaliplatin, leucovorin calcium, and fluorouracil as in arm A. Treatment repeats every 14 days for up to 12 courses in the absence of unacceptable toxicity or recurrent disease.
  oxaliplatin: Given IV
  leucovorin calcium: Given IV
  fluorouracil: Given IV
  cetuximab: Given IV
- Arm E (Combination Chemotherapy, Monoclonal Antibody): Patients receive cetuximab as in arm D and irinotecan, leucovorin calcium, and fluorouracil as in arm B. Treatment repeats every 14 days for up to 12 courses in the absence of unacceptable toxicity or recurrent disease.
  irinotecan hydrochloride: Given IV
  leucovorin calcium: Given IV
  fluorouracil: Given IV
  cetuximab: Given IV
- Arm F (Combination Chemotherapy, Monoclonal Antibody): Patients receive cetuximab as in arm D and chemotherapy as in arm C.
  irinotecan hydrochloride: Given IV
  oxaliplatin: Given IV
  leucovorin calcium: Given IV
  fluorouracil: Given IV
  cetuximab: Given IV
- Arm G (Locally Directed Therapy): Patients determined to have mutated KRAS (or KRAS not evaluable) will be assigned to an event monitoring arm in which adjuvant therapy will be determined and assigned by the treating oncologist. The determination of the type of therapy, duration of treatment, and dose modification will be the responsibility of the treating oncologists.
  Locally Directed Therapy: Patients determined to have mutated KRAS (or KRAS not evaluable) will be assigned to an event monitoring arm in which adjuvant therapy will be determined and assigned by the treating oncologist. The determination of the type of therapy, duration of treatment, and dose modification will be the responsibility of the treating oncologists.
Arm/Group | Arm A (Combination Chemotherapy) | Arm B (Combination Chemotherapy) | Arm C (Combination Chemotherapy) | Arm D (Combination Chemotherapy, Monoclonal Antibody) | Arm E (Combination Chemotherapy, Monoclonal Antibody) | Arm F (Combination Chemotherapy, Monoclonal Antibody) | Arm G (Locally Directed Therapy)
Serious Adverse Events (participants affected / at risk) | 93/1378 | 9/108 | 11/108 | 150/1326 | 4/42 | 5/44 | 0/0
Other Adverse Events (participants affected / at risk) | 688/1378 | 53/108 | 60/108 | 928/1326 | 26/42 | 33/44 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Combination Chemotherapy) (N=1378) | Arm B (Combination Chemotherapy) (N=108) | Arm C (Combination Chemotherapy) (N=108) | Arm D (Combination Chemotherapy, Monoclonal Antibody) (N=1326) | Arm E (Combination Chemotherapy, Monoclonal Antibody) (N=42) | Arm F (Combination Chemotherapy, Monoclonal Antibody) (N=44) | Arm G (Locally Directed Therapy) (N=0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asystole (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Cardiopulmonary arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischemia (Cardiac disorders) | 6 (7) | 0 (0) | 1 (1) | 9 (9) | 1 (1) | 0 (0) | 0 (0)
Premature ventricular contractions (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Colonic fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Colonic stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 15 (15) | 0 (0) | 1 (1) | 20 (20) | 0 (0) | 0 (0) | 0 (0)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endoscopy small intestine abnormal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Esophageal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Esophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 1 (1) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gallbladder pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatobiliary disease (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 6 (6) | 0 (0) | 0 (0) | 17 (17) | 0 (0) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infectious colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infectious meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 7 (7) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Cardiac troponin T increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INR increased (Investigations) | 4 (5) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 13 (15) | 1 (1) | 1 (1) | 8 (8) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 7 (7) | 1 (1) | 2 (2) | 10 (10) | 0 (0) | 1 (1) | 0 (0)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Serum glucose decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Serum magnesium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 10 (10) | 0 (0) | 0 (0) | 20 (20) | 0 (0) | 0 (0) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 6 (6) | 0 (0) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder hemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2) | 6 (6) | 2 (2) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Masculinization (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 5 (5) | 2 (2) | 0 (0) | 9 (9) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Combination Chemotherapy) (N=1378) | Arm B (Combination Chemotherapy) (N=108) | Arm C (Combination Chemotherapy) (N=108) | Arm D (Combination Chemotherapy, Monoclonal Antibody) (N=1326) | Arm E (Combination Chemotherapy, Monoclonal Antibody) (N=42) | Arm F (Combination Chemotherapy, Monoclonal Antibody) (N=44) | Arm G (Locally Directed Therapy) (N=0)
Febrile neutropenia (Blood and lymphatic system disorders) | 12 (12) | 2 (3) | 3 (3) | 30 (33) | 1 (1) | 1 (1) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 6 (9) | 0 (0) | 0 (0) | 8 (11) | 0 (0) | 0 (0) | 0 (0)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Asystole (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 2 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cardiac pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conduction disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Premature ventricular contractions (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Eyelid function disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Watering eyes (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 31 (32) | 1 (1) | 2 (2) | 28 (35) | 1 (1) | 3 (5) | 0 (0)
Anal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Cecal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 9 (10) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 107 (125) | 15 (28) | 13 (17) | 192 (250) | 6 (7) | 7 (11) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 18 (20) | 2 (2) | 2 (2) | 63 (77) | 3 (4) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Ileal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 1 (2) | 0 (0)
Intestinal necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 18 (19) | 2 (2) | 2 (6) | 44 (51) | 3 (3) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 35 (41) | 9 (10) | 6 (6) | 56 (66) | 0 (0) | 8 (10) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 5 (6) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 40 (44) | 7 (10) | 5 (5) | 41 (45) | 0 (0) | 4 (6) | 0 (0)
Chest pain (General disorders) | 5 (6) | 1 (1) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 53 (80) | 2 (2) | 9 (11) | 77 (122) | 1 (1) | 2 (2) | 0 (0)
Flu-like symptoms (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait abnormal (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General symptom (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ill-defined disorder (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 4 (5) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatobiliary disease (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 28 (29) | 0 (0) | 2 (2) | 62 (65) | 1 (2) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 5 (5) | 0 (0) | 1 (2) | 13 (14) | 1 (1) | 1 (1) | 0 (0)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ileal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 5 (5) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Infectious colitis (Infections and infestations) | 8 (10) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Joint infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 10 (10) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 1 (1) | 0 (0)
Salivary gland infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 4 (4) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 3 (4) | 1 (1) | 0 (0) | 24 (41) | 1 (1) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper aerodigestive tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (4) | 0 (0) | 0 (0) | 8 (8) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arterial injury - Extremity-lower (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injury to superior vena cava (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal stoma site bleeding (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 22 (33) | 3 (3) | 5 (8) | 18 (34) | 1 (1) | 2 (2) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (2) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 16 (21) | 1 (1) | 0 (0) | 14 (18) | 1 (1) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 10 (10) | 0 (0) | 0 (0) | 11 (12) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coagulopathy (Investigations) | 3 (7) | 0 (0) | 0 (0) | 3 (10) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 2 (5) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
INR increased (Investigations) | 16 (39) | 0 (0) | 1 (3) | 15 (30) | 0 (0) | 0 (0) | 0 (0)
Leukocyte count decreased (Investigations) | 25 (32) | 1 (1) | 0 (0) | 31 (36) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 5 (6) | 0 (0) | 1 (1) | 8 (14) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 131 (148) | 14 (18) | 18 (20) | 154 (175) | 3 (4) | 4 (4) | 0 (0)
Platelet count decreased (Investigations) | 6 (6) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Serum cholesterol increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight gain (Investigations) | 1 (1) | 1 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 2 (3) | 0 (0) | 0 (0) | 9 (18) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 9 (9) | 1 (1) | 0 (0) | 28 (35) | 1 (1) | 2 (3) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 42 (99) | 8 (37) | 6 (12) | 32 (69) | 1 (2) | 1 (6) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 10 (10) | 1 (1) | 3 (3) | 39 (42) | 0 (0) | 1 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Serum albumin decreased (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0) | 8 (11) | 0 (0) | 0 (0) | 0 (0)
Serum calcium decreased (Metabolism and nutrition disorders) | 6 (6) | 0 (0) | 1 (1) | 9 (9) | 0 (0) | 1 (1) | 0 (0)
Serum magnesium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 26 (43) | 0 (0) | 2 (4) | 0 (0)
Serum magnesium increased (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0) | 9 (13) | 0 (0) | 1 (2) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 33 (43) | 2 (3) | 1 (1) | 84 (120) | 0 (0) | 2 (2) | 0 (0)
Serum potassium increased (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 4 (5) | 0 (0) | 0 (0) | 9 (12) | 0 (0) | 0 (0) | 0 (0)
Serum triglycerides increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acoustic nerve disorder NOS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 12 (14) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (8) | 0 (0) | 2 (3) | 10 (12) | 0 (0) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Laryngeal (Nervous system disorders) | 7 (11) | 1 (1) | 3 (7) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Neurological disorder NOS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Paresthesias (Nervous system disorders) | 169 (295) | 0 (0) | 3 (3) | 121 (220) | 4 (7) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 6 (10) | 0 (0) | 1 (1) | 10 (14) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 67 (116) | 2 (2) | 0 (0) | 67 (109) | 1 (1) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 5 (5) | 1 (1) | 0 (0) | 8 (10) | 0 (0) | 0 (0) | 0 (0)
Syncope vasovagal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Trigeminal nerve disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vagus nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (6) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 2 (3) | 0 (0) | 1 (1) | 4 (7) | 0 (0) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Kidney pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irregular menstruation (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 0 (0) | 1 (1) | 12 (18) | 0 (0) | 2 (3) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 13 (18) | 2 (2) | 0 (0) | 28 (32) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 8 (9) | 0 (0) | 2 (2) | 0 (0)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 2 (2) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 11 (15) | 1 (1) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 16 (19) | 2 (2) | 0 (0) | 40 (56) | 1 (1) | 2 (2) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 24 (38) | 2 (3) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 156 (259) | 7 (11) | 7 (12) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 1 (1) | 116 (194) | 4 (8) | 8 (12) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 7 (9) | 0 (0) | 0 (0) | 4 (7) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 43 (74) | 3 (3) | 5 (5) | 49 (69) | 2 (2) | 0 (0) | 0 (0)
Vascular disorder (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Accrual to arms A and D terminated early based on the results of the planned 2nd interim analysis. Sample sizes limit statistical conclusions for data from the irinotecan treated patients as those treatment arms were discontinued early in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less